CLINICAL TRIAL: NCT05971446
Title: Visual Function as a Novel Outcome Measure Following Neonatal Hypoxic Ischemic Encephalopathy
Brief Title: Healthy Little Eyes
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Meriter Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1243; SMPH\PEDIATRICS\PICU (Other: UW Madison); Protocol Version 4/11/2025 (Other: UW Madison)
Record Dates: First submitted 2023-06-27; First posted 2023-08-02 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Neonatal Encephalopathy; Encephalopathy
Keywords: neonatal; visual evoked potential; electroretinogram
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Brain Diseases | interventions — Electroretinography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Participants with HIE
  Interventions: Device: Visual Evoked Potential (VEP); Device: Electroretinogram (ERG)
- Healthy participants
  Interventions: Device: Visual Evoked Potential (VEP); Device: Electroretinogram (ERG)

INTERVENTIONS:
Device: Visual Evoked Potential (VEP) — Small gold-cup electrodes will be placed on the participant's head using a small dot of adhesive paste. The handheld device is then connected to the electrodes, and the participant's eyes are exposed to a light flicker. Each eye will be tested separately, and while testing one eye, the other eye may be patched.
Device: Electroretinogram (ERG) — Skin electrodes will be placed under each eye. Eyes will then be exposed to a flashing light. Each eye will be tested separately and while testing one eye, the other eye may be patched.

SUMMARY:
The purpose of this research study is to gather more information on how eye injury is related to a baby's future development and see if eye function and brain test results can be used, along with current measures, to better diagnose and treat babies with hypoxic-ischemic encephalopathy (HIE).

Participants will undergo up to two eye exam sessions, involving both Visual Evoked Potential (VEP) and Electroretinogram (ERG) exams.

DETAILED DESCRIPTION:
Specific Aims/Study Objectives:

In this proposed longitudinal study, the investigators hypothesize that the early visual function findings will correlate with the neurodevelopmental and neuroimaging outcomes in children who sustain HIE. The investigators will test this hypothesis through the following specific aims:

* Specific Aim 1 will determine the correlation of the ERG results as a measure of the retinal function obtained at around birth, 3, 9, 18 or 30 months of life and neurodevelopmental-neuroimaging outcomes from birth through 36 months.
* Specific Aim 2 will determine the correlation of the VEP as a measure of the visual cortical function obtained at around birth, 3, 9, 18 or 30 months of life and neurodevelopmental-neuroimaging outcomes from birth through 36 months.
* Specific Aim 3 will collect ERG and VEP results from well babies in the Newborn Nursery and compare results to neonates with HIE.
* Specific Aim 4 will determine if machine learning will predict the clinical outcomes using VEP, ERG, and EEG waveform data, as well as MR imaging files (exploratory)

As health care providers, the investigators' goal is to develop a noninvasive and novel quantitative tool to improve the neurodevelopmental outcome of neonates and to support them in attaining maximum functional potential in childhood and beyond.

ELIGIBILITY:
HIE Neonate Inclusion Criteria:

* Inpatient Neonates diagnosed with HIE
* Pediatric patients who are less than 78 hours of age at the time of enrollment
* Participants whose parent/legal guardian is able to complete consenting process in English

HIE Neonate Exclusion Criteria:

* Participants with prenatally diagnosed or congenital brain and/or eye abnormalities not associated with HIE, including but not limited to microphthalmia, anophthalmia, congenital cataract, eye or eyelid coloboma, congenital glaucoma, CMV retinitis, optic nerve hypoplasia, aniridia, cryptophthalmos, globe abnormalities
* Participants who have a known central nervous system illness other than HIE, including but not limited to congenital brain malformations or congenital hydrocephalus
* Participants whose parent/legal guardian is unable to provide informed consent, including participants who are in foster care, participants within state custody, and participants of minor parents

Waisman, AFCH NBFU, or CERU Clinic HIE Patient Inclusion Criteria:

* Pediatric patients who have a diagnosis of HIE and present to the Newborn Follow Up Clinic
* Pediatric patients who are less than 36 months of age at the time of enrollment
* Participants whose parent/legal guardian is able to complete consenting process in English

Waisman, AFCH NBFU, or CERU Clinic HIE Patient Exclusion Criteria:

* Participants with prenatally diagnosed or congenital brain and/or eye abnormalities not associated with HIE, including but not limited to microphthalmia, anophthalmia, congenital cataract, eye or eyelid coloboma, congenital glaucoma, CMV retinitis, optic nerve hypoplasia, aniridia, cryptophthalmos, globe abnormalities
* Participants who have a known central nervous system illness not associated with HIE and its complications. Complications may include seizures, hydrocephalus, and stroke, which are NOT exclusionary. Examples of exclusionary conditions include but are not limited to traumatic brain injury outside the perinatal period, meningitis, or diagnosis of brain tumor
* Participants whose parent/legal guardian is unable to provide informed consent, including participants who are in foster care, participants within state custody, and participants of minor parents

Well Baby Inclusion Criteria:

* Patient in Meriter's Newborn Nursery
* ≥37 and <42 weeks gestational age
* 5-minute Apgar Score ≥7
* Occipital Frontal Circumference (OFC) is within average limits for age (<97th percentile and >3rd percentile)

Well Baby Exclusion Criteria:

* Admitted to the NICU for any reason
* Known genetic abnormality
* Diagnosed with HIE
* Diagnosed with Hypoglycemia
* Diagnosed with Hyperbilirubinemia requiring phototherapy
* Identified prenatal exposure to substances, including illicit drugs, alcohol, and/or tobacco
* Known or suspected neonatal infection requiring treatment (e.g., antibiotics)
* TORCH infections
* Abnormal newborn hearing screen
* Abnormal toxicology screening
* Identified as large for gestational age (LGA) or small for gestational age (SGA)
* Participants with prenatally diagnosed or congenital eye abnormalities, including but not limited to microphthalmia, anophthalmia, congenital cataract, eye or eyelid coloboma, congenital glaucoma, CMV retinitis, optic nerve hypoplasia, aniridia, cryptophthalmos, globe abnormalities, and nystagmus
* Subjects who have a known central nervous system illness or malformation, including but not limited to congenital brain malformations or congenital hydrocephalus
* Participants whose parent/legal guardian is unable to provide informed consent, including subjects who are in foster care, subjects within state custody, and subjects of minor parents
* The attending medical team does not approve

Max Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. HIE Neonates in the NICU at AFCH or Meriter who are less than 78 hours old
  2. HIE Neonates at Waisman, AFCH Newborn Follow-up Clinic, or CERU Clinic who are less than 78 hours old
  3. Well babies at the Meriter Newborn Nursery who are less than 36 months of age
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the correlation between retinal function and neurodevelopmental outcomes | Through 30 months of life
  The least absolute shrinkage and selection operator technique will be utilized to determine whether ERG measures predict neurodevelopmental outcomes
To evaluate the correlation between retinal function and neuroimaging outcomes | Within first 5 days of life
  The least absolute shrinkage and selection operator technique will be utilized to determine whether ERG measures predict neuroimaging outcomes
To evaluate the correlation between visual cortical function and neurodevelopmental outcomes | Through 30 months of life
  The least absolute shrinkage and selection operator technique will be utilized to determine whether VEP measures predict neurodevelopmental outcomes
To evaluate the correlation between visual cortical function and neuroimaging outcomes | Within first 5 days of life
  The least absolute shrinkage and selection operator technique will be utilized to determine whether VEP measures predict neuroimaging outcomes
Compare ERG results between healthy babies and babies with HIE | Within first 5 days of life
  The ERG results from healthy babies will be compared to those of babies with HIE
Report Shape of the VEP results for healthy babies and babies with HIE | Within first 5 days of life
  The shape of the waveform will be reported as a categorical variable: sharp, slanted, blunt, or multiple peaks
Compare Amplitude of the VEP results between healthy babies and babies with HIE | Within first 5 days of life
  The amplitude will be reported as differences in microvolt responses between groups.
Compare Latency of the VEP results between healthy babies and babies with HIE | Within first 5 days of life
  The latency will be reported as differences in timing (measured in milliseconds) between groups.
Compare Transocular Shape, Amplitude, and Latency Difference of the VEP results between healthy babies and babies with HIE | Within first 5 days of life
  The Transocular Shape Difference will be reported as differences in shape between the two eyes compared across groups, reported as a categorical variable: sharp, slanted, blunt, or multiple peaks.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Cengiz, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No